CLINICAL TRIAL: NCT00183521
Title: Respiratory Therapeutic Procedures in Panic Disorder
Brief Title: Breathing Regulation Training for Individuals With Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Walton T Roth, M.D., Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH066953 (NIH); R01MH066953 (NIH); DATR A2-AIR
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Panic Disorder
Keywords: Hyperventilation; Breathing Exercises; Carbon Dioxide; Panic Attack
MeSH Terms: conditions — Panic Disorder; Hyperventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive raise-CO2 breathing regulation training
  Interventions: Behavioral: Raise-CO2 breathing regulation training
- 2 (Experimental): Participants will receive lower-CO2 breathing regulation training
  Interventions: Behavioral: Lower-CO2 breathing regulation training
- 3 (Active Comparator): Participants will receive no breathing regulation training
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Raise-CO2 breathing regulation training — Reverse hyperventilation (defined by low arterial CO2) is often characteristic of individuals with panic disorder. Participants will be randomly assigned to one of three groups: raise-CO2 breathing, lower-CO2 breathing, or a control group. Participants in the raise-CO2 group will be taught techniques to recover from hyperventilation faster.
  Arms: 1
Behavioral: Lower-CO2 breathing regulation training — According to the false suffocation alarm theory, anxiety is experienced when an overly sensitive hypothalamic mechanism is triggered by rising pCO2. Participants in the lower-CO2 group will be taught techniques to reach hyperventilation levels, then switch to breathing techniques that reduce hyperventilation symptoms.
  Arms: 2
Behavioral: Control — Participants in the control group will not be taught any breathing techniques but will be included in all assessments.
  Arms: 3

SUMMARY:
This study will compare two different breathing regulation techniques to determine which is more effective in reducing the rate of panic attacks in people with panic disorder.

DETAILED DESCRIPTION:
PD is a serious condition characterized by episodes of rapid heart rate, difficulty breathing, and other symptoms of fear. Explanations for panic attacks have been proposed in two theories: suffocation alarm theory and hyperventilation theory. The suffocation alarm theory claims that panic attacks are due to a "suffocation monitor" in the brain, erroneously signaling a lack of useful air. The hyperventilation theory suggests that stressful events cause people to slightly hyperventilate; some people have panic attacks as a result of their overreaction to the dizziness and lightheadedness they feel from hyperventilation. Both theories note the role of carbon dioxide (CO2) in panic attacks; they suggest that rising CO2 levels in arterial blood act as a panic stimulus. This study will compare two types of breathing regulation techniques based on the panic attack theories to determine which is more effective in reducing panic symptoms in people with PD.

This study will last 4 weeks and will include both people with PD and those without the condition. Participants will be randomly assigned to one of three groups: raise-CO2 breathing, lower-CO2 breathing, or a control group. Participants in both the raise-CO2 and lower-CO2 breathing groups will have five sessions of training in which they will learn specific breathing techniques. Participants in the raise-CO2 group will be taught techniques to recover from hyperventilation faster; participants in the lower-CO2 group will be taught techniques to reach hyperventilation levels, then switch to breathing techniques that reduce hyperventilation symptoms. Participants in the control group will not be taught any breathing techniques but will be included in all assessments.

Participants will be assessed at study entry, during each breathing training session, and at Months 1 and 6 after the study. During each assessment, questionnaires and self-report scales will be used to measure cognitive, psychological, and physiological changes related to participants' breathing.

ELIGIBILITY:
Inclusion Criteria for Participants With PD:

* Diagnosis of PD
* History of panic attacks that are at least moderately severe in frequency and severity
* Able and willing to comply with all study requirements

Exclusion Criteria for All Participants:

* History of chest pain, heart attack, congestive heart failure, or clinically significant irregular heartbeat
* History of blood circulation problems or cerebrovascular accidents
* Diabetes mellitus
* Asthma or chronic obstructive pulmonary disease (COPD)
* History of schizophrenia, bipolar disorder, or dementia
* Drugs which would affect breathing
* Alcohol or other substance abuse within 1 year prior to study entry
* Current use of any recreational drugs or consumption of more than 15 alcoholic drinks per week

Exclusion Criteria for Participants Without PD:

* History of anxiety disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2005-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Breathing regulation | Measured at Month 6 after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Walton T. Roth, MD, Principal Investigator — Stanford University and VA Health Care System
Locations (1):
- Stanford University & VA Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Kim S, Wollburg E, Roth WT. Opposing breathing therapies for panic disorder: a randomized controlled trial of lowering vs raising end-tidal P(CO(2)). J Clin Psychiatry. 2012 Jul;73(7):931-9. doi: 10.4088/JCP.11m07068. PMID 22901344